CLINICAL TRIAL: NCT01259427
Title: Reducing Internalized Stigma In People With Serious Mental Illness
Acronym: ESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 09-340
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression With Psychotic Features
Keywords: Mental Disorders; Psychotic Disorders; Schizophrenia; Stigmatization; Mood Disorders; Schizophrenia and Disorders with Psychotic Feature
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders; Stereotyping; Mood Disorders | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Ending Self Stigma (Experimental): Ending Self Stigma (ESS): Ending Self Stigma (ESS) is a 9-session small-group (4-8 persons) course designed to help individuals with serious mental Illness (SMI) develop skills to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes. Sessions combine in-class lecture, discussion of relevance to group members' personal experiences, review and practice of strategies and skills, and group sharing, support, and problem-solving. Each session is designed to focus on a specific strategy for addressing self-stigma.
  Interventions: Behavioral: Ending Self Stigma (ESS)
- Arm 2: Health and Wellness Group (Active Comparator): Health and Wellness Group: The Health and Wellness group is a 9-session small-group (4-8 persons) course designed for individuals with serious mental illness (SMI). Each session focuses on discussion of specific health and wellness related issues and education on ways to better manage health related concerns (e.g., physical activity/exercise, nutrition, managing fatigue/sleep, tobacco and other substance use, etc).
  Interventions: Behavioral: Health and Wellness Group

INTERVENTIONS:
Behavioral: Ending Self Stigma (ESS) — Ending Self Stigma (ESS) is a 9-session small-group (4-8 persons) course designed to help individuals with serious mental Illness (SMI) develop skills to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes. Sessions combine in-class lecture, discussion of relevance to group members' personal experiences, review and practice of strategies and skills, and group sharing, support, and problem-solving. Each session is designed to focus on a specific strategy for addressing self-stigma.
  Arms: Arm 1: Ending Self Stigma
Behavioral: Health and Wellness Group — The Health and Wellness group is a 9-session small-group (4-8 persons) course designed for individuals with serious mental illness (SMI). Each session focuses on discussion of specific health and wellness related issues and education on ways to better manage health related concerns (e.g., physical activity/exercise, nutrition, managing fatigue/sleep, tobacco and other substance use, etc).
  Arms: Arm 2: Health and Wellness Group

SUMMARY:
The purpose of this study is to determine if Ending Self-Stigma (ESS), a 9-session group intervention designed to assist veterans with serious mental illness to develop skills (SMI) to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes, is more effective in reducing internalized stigma and its associated effects than an active comparison group.

DETAILED DESCRIPTION:
Background:

Stigmatizing beliefs and attitudes about mental illness are prevalent and exposure to stigma is common among people with mental illness. The negative effects of stigma are compounded when a veteran with Serious Mental Illness (SMI) internalizes these stigmatizing assumptions and stereotypes. Internalized stigma refers to the process in which a person with mental illness cognitively or emotionally absorbs negative messages or stereotypes about mental illness and comes to believe them and apply them to him/herself. Internalized stigma is evident among veterans with SMI and can lead to decreased self-efficacy, increased depression, social withdrawal, and curtailed pursuit of recovery goals.

Objectives:

The investigators developed Ending Self Stigma (ESS), a 9-session group intervention to assist veterans with SMI to develop skills to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes. The primary objectives of this project are to compare the effects of ESS to a general health and wellness group in: 1) reducing internalized stigma and 2) improving proximal psychosocial outcomes (e.g., self-efficacy, belonging, recovery orientation). Secondary objectives include assessing the effects of ESS on improving distal psychosocial outcomes (e.g., quality of life, social functioning) and examining if improvements are maintained 6-months post-treatment.

Methods:

This study is a randomized trial of veterans with SMI receiving outpatient mental health services from three VA Medical Centers. Participants are randomly assigned to ESS or a general health and wellness group, which they attend once a week for 9 weeks. ESS focuses on teaching strategies/tools to help participants address self-stigma. The health and wellness group focuses on providing information/ education to help participants better manage health-related concerns (e.g. physical activity, nutrition). Participants complete assessments at baseline, post-treatment, and 6-months post-treatment. A two-level mixed effects model with adjustment for baseline response will be used to address the primary and secondary aims. Qualitative data on veterans' experiences of and strategies for coping with internalized stigma are being collected from a subset of veterans from both conditions to compare experiences of veterans in both groups and explore any reasons for ESS drop-out.

Status:

Data collection for the project is completed. Analysis of 6-month post-treatment assessments and qualitative interviews are currently being conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* Schizoaffective disorder
* Bipolar Disorder
* or Major Depression with Psychotic Features
* Age 18 to 80
* Receiving services at one of VA Medical Center study sites
* Ability and willingness to provide consent to participate
* Agreement obtained from the treating clinician that the patient is clinically stable enough to participate in the study

Exclusion Criteria:

* Severe or profound mental retardation by chart review

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drapalski, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (3):
- United States (3):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Perry Point VA Medical Center VA Maryland Health Care System, Perry Point, MD, Perry Point, Maryland

REFERENCES:
- [Result] Yanos PT, Lucksted A, Drapalski AL, Roe D, Lysaker P. Interventions targeting mental health self-stigma: A review and comparison. Psychiatr Rehabil J. 2015 Jun;38(2):171-178. doi: 10.1037/prj0000100. Epub 2014 Oct 13. PMID 25313530
- [Derived] Drapalski AL, Tonge N, Muralidharan A, Brown CH, Lucksted A. Even mild internalized stigma merits attention among adults with serious mental illness. Psychol Serv. 2023;20(Suppl 2):166-174. doi: 10.1037/ser0000744. Epub 2023 Mar 9. PMID 36892916
- [Derived] Drapalski AL, Lucksted A, Brown CH, Fang LJ. Outcomes of Ending Self-Stigma, a Group Intervention to Reduce Internalized Stigma, Among Individuals With Serious Mental Illness. Psychiatr Serv. 2021 Feb 1;72(2):136-142. doi: 10.1176/appi.ps.201900296. Epub 2020 Nov 25. PMID 33234053
- [Derived] Wastler H, Lucksted A, Phalen P, Drapalski A. Internalized stigma, sense of belonging, and suicidal ideation among veterans with serious mental illness. Psychiatr Rehabil J. 2020 Jun;43(2):91-96. doi: 10.1037/prj0000386. Epub 2019 Aug 15. PMID 31414842
- [Derived] Jahn DR, Leith J, Muralidharan A, Brown CH, Drapalski AL, Hack S, Lucksted A. The influence of experiences of stigma on recovery: Mediating roles of internalized stigma, self-esteem, and self-efficacy. Psychiatr Rehabil J. 2020 Jun;43(2):97-105. doi: 10.1037/prj0000377. Epub 2019 Jun 24. PMID 31233321

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were consented but indicated that they were unable to continue their participation prior to completing the baseline assessment. One participant was determined to be ineligible after randomization and was withdrawn from the study.
Groups:
- Arm 2: Health and Wellness Group: Health and Wellness Group: The Health and Wellness group is a 9-session small-group (4-8 persons) course designed for individuals with serious mental illness (SMI). Each session focuses on discussion of specific health and wellness related issues and education on ways to better manage health related concerns (e.g., physical activity/exercise, nutrition, managing fatigue/sleep, tobacco and other substance use, etc.).
Period: Overall Study
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Started | 124 | 124
Completed | 106 | 110
Not Completed | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.8) | 53.3 (9.5) | 53.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 108 | 107 | 215

OUTCOME MEASURES:

1. Primary Outcome: Internalized Stigma of Mental Illness Inventory (Internalized Stigma)
Description: The Internalized Stigma of Mental Illness Inventory was used to measure of internalized or self-stigma. A total score is calculated by taking an average of the responses on the items (range=1 to 4). Higher total scores indicate greater internalized stigma.
Time Frame: ~3 months (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline | 2.2 (.4) | 2.2 (.4)
  Post Treatment | 2.1 (.4) | 2.1 (.5)

2. Primary Outcome: Maryland Assessment of Recovery for Serious Mental Illness Scale (Recovery)
Description: The Maryland Assessment of Recovery in Serious Mental Illness is a self-report measure of recovery in people with serious mental illness. A total score was calculated by summing item responses (range=25 to 125), with higher total scores indicating greater self-reported recovery.
Time Frame: ~3 1/2 months (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline | 94.9 (18.1) | 95.7 (18.0)
  Post-treatment | 96.7 (16.4) | 97.3 (18.4)

3. Primary Outcome: General Self-Efficacy Scale
Description: The General Self-efficacy measure was used to measure of self-efficacy. A total score was calculated by averaging the responses on the items (range=1 to 5), with higher scores indicating greater self-efficacy.
Time Frame: ~3 1/2 months (post-treatment)
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
unit on a scale
  Baseline | 3.6 (.7) | 3.5 (.8)
  Post-treatment | 3.6 (.7) | 3.7 (.7)

4. Primary Outcome: Sense of Belonging Instrument (Belonging)
Description: The Sense of Belonging Instrument was used to measure perceived belongingness. The measure includes two subscales: the psychological experience of belonging (SOBI-P) and antecedents that foster belonging (SOBI-A). An average of the sum of the items in each subscale were used to calculate the total score for that subscale. The total score of the SOBI-P ranges from 18 to 72, with higher scores indicating less experienced belonging. The total score of the SOBI-A ranges from 14-56 with higher score indicating greater antecedents that foster belonging.
Time Frame: ~3 1/2 months (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline: SOBI-P | 40.4 (5.5) | 39.7 (6.1)
  Post-Treatment: SOBI-P | 39.6 (5.8) | 39.9 (5.4)
  Baseline: SOBI-A | 46.6 (10.2) | 46.0 (11.4)
  Post-Treatment: SOBI-A | 47.8 (9.6) | 48.8 (11.2)

5. Secondary Outcome: Quality of Life
Description: The Satisfaction with Life in General item from the Brief Quality of Life Scale was used to assess self-reported life satisfaction. The item is rated on a 7-point scale that ranges from terrible to delighted (range=1 to 7), with greater scores indicating more satisfaction.
Time Frame: ~3 1/2 months (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline | 4.3 (1.3) | 4.4 (1.5)
  Post-treatment | 4.6 (1.3) | 4.7 (1.4)

6. Secondary Outcome: Social Engagement/Withdrawal
Description: The total score of the Social Engagement/Withdrawal subscale of the Social Functioning Scale was used to measure social engagement. The total score ranges from 0 to 15 with higher scores indicating greater social engagement.
Time Frame: ~3 1/2 months (post-treatment)
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Number analyzed (Participants) | 124 | 124
unit on a scale
  Baseline | 9.6 (2.5) | 9.5 (2.3)
  Post-treatment | 9.7 (2.4) | 10.0 (2.5)

ADVERSE EVENTS:
Time Frame: Duration of participants involvement in the study, up to ~11 months
Arm/Group | Arm 1: Ending Self Stigma | Arm 2: Health and Wellness Group
Serious Adverse Events (participants affected / at risk) | 7/124 | 7/124
Other Adverse Events (participants affected / at risk) | 0/124 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Ending Self Stigma (N=124) | Arm 2: Health and Wellness Group (N=124)
Psychiatric hospitalization (Psychiatric disorders) | 5 (5) | 5 (5) — All psychiatric hospitalizations that occurred during the study were reported to the local IRB and unrelated to study participation
Death (General disorders) | 1 (1) | 2 (2) — All deaths that occurred during the study were reported to the local IRB and were determined to be unrelated to study participation
Medical Hospitalization (General disorders) | 1 (1) | 0 (0) — All medical hospitalizations that occurred during the study were reported to the local IRB and unrelated to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes